CLINICAL TRIAL: NCT05728801
Title: Decoding the Cognitive Trajectory of Hong Kong SuperAgers: a Longitudinal Follow-up Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, LU Hanna, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: 2019.078
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Age-related Cognitive Decline; Cognitive Deterioration; Dementia, Mild
Keywords: Cognitive maintenance; Cognitive ageing; Superagers; Cognition; Quality of life; Brain health
MeSH Terms: conditions — Dementia; Lymphoma, Follicular | interventions — Aging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Superagers: SuperAgers are determined by the scores of global cognitive function. This ensured that the participants are divided by a measure relevant to the current study without directly biasing the results toward the domain of interest.
  Interventions: Diagnostic Test: Ageing
- Normal ageing elderly: The cases with the scores of cognitive performance within 1.5 standard deviation (SD) of age and education matched normative values derived from our cohort study, of which presented with HK MoCA score greater than 26 and CDR score equal to 0
  Interventions: Diagnostic Test: Ageing
- Neurocognitive disorders patients: NCD patients are deﬁned as: evidence of modest decline in one or more cognitive domains, which is set as ≥ 1.5 SD below the age- and education-adjusted normative scores; no interference with independence in everyday activities; and no comorbid major psychiatric disorders.
  Interventions: Diagnostic Test: Ageing

INTERVENTIONS:
Diagnostic Test: Ageing — Using comprehensive cognitive tests to quality the domain-specific cognitive changes during ageing.

SUMMARY:
This is a prospective follow-up study conducted at the Department of Psychiatry, The Chinese University of Hong Kong. The participants, including high-performing elderly (SuperAgers), normal ageing elderly and neurocognitive disorder (NCD) patients will be re-invited from our previous cohort (2013-2014) (N=488).

DETAILED DESCRIPTION:
Objectives: This study aims to investigate the cognitive changes in older adults with different cognitive statuses.

ELIGIBILITY:
Inclusion Criteria:

* SuperAgers are determined by the scores of global cognitive function. This ensured that the participants are divided by a measure relevant to the current study without directly biasing the results toward the domain of interest;
* Normal aging: the cases with the scores of cognitive performance within 1.5 standard deviation (SD) of age and education matched normative values derived from our cohort study, of which presented with HK MoCA score greater than 26 and CDR score equal to 0;
* NCD patients are deﬁned as: evidence of modest decline in one or more cognitive domains, which is set as ≥ 1.5 SD below the age- and education-adjusted normative scores; no interference with independence in everyday activities; and no comorbid major psychiatric disorders.

Exclusion Criteria:

* History of bipolar disorders or psychosis;
* History of major neurological deﬁcits including stroke, transient ischemic attack or traumatic brain injury;
* Comorbidities with depressive symptoms.

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: High-performing elderly (SuperAgers) and the cases with normal ageing and neurocognitive disorder (NCD) will be re-invited in this study.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Global cognition will be measured by the Montreal Cognitive Assessment Hong Kong version (HK MoCA) | 2022-2024
  The Montreal Cognitive Assessment Hong Kong version (HK MoCA) is a validated and widely used screening assessment for detecting cognitive impairment, which measures an array of cognitive functions such as visuospatial, memory, language and attention.HK MoCA score less than 26 indicates cognitive impairments.
Complex attention will be measured by Attention Network Test (ANT) | 2022-2024
  Attention Network Test (ANT). The ANT paradigm (Download from: https://www.sacklerinstitute.org/cornell/assays_and_tools/ant/jin.fan/), as a computerized test, was used and performed by E-Prime 3.0 (Psychology Software Tools, PA, USA). Within ANT paradigm, there are four types of cue: no cue, center cue, double cue, and spatial cue; and three types of ﬂanker: neutral, congruent, and incongruent. In a given trial, a central cross-ﬁxation point presents for 400 to 1,600 ms (randomized), subsequently is replaced for 100 ms by one of four warning cues. The target, a central arrow could appear above or below the cross-ﬁxation and is surrounded by two ﬂankers on each side.

SECONDARY OUTCOMES:
Learning and memory will be measured by Word list learning test (WLLT) | 2022-2024
  Word list learning test (WLLT) consisting of fifteen semantically non-associated words that is presented consecutively over three free trials of immediate recall (i.e., learning ability), a 20-min delayed recall (to prevent recency effects) and followed by yes/no recognition (i.e., recognition memory). Based on the proxies we developed in our previous work, components of learning and memory function will be evaluated and compared across groups, including working memory capacity (WMC), forgetting rate, delayed recall, initial learning, best learning, learning over trials (LOT) and learning ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Hanna LU, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Tai Po Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Hong Kong SuperAgers — https://www.psychiatry.cuhk.edu.hk/members/dr-hanna-lu/